CLINICAL TRIAL: NCT00390962
Title: Copeptin as a Novel Diagnostic and Prognostic Marker in the Management of Neurological and Neurosurgical Patients With Sodium Imbalance The "COSMOS"-Study (Copeptin in Osmoregulation and Stress Assessment)
Brief Title: The "COSMOS"-Study (Copeptin in Osmoregulation and Stress Assessment)
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Other Study IDs: EKBB 157/06
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: copeptin; vasopressin; Adh; SIADH; diabetes insipidus; stroke; risk factors; Neurological patients with ischemic and hemorrhagic stroke and patients undergoing intracranial surgery.
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Diabetes Insipidus; Carcinoma, Intraductal, Noninfiltrating; Inappropriate ADH Syndrome; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bood sampling

SUMMARY:
Sodium imbalance is common and an adverse prognostic factor in hospitalized patients. However, identifying the causes of sodium imbalance is challenging in clinical practice. Levels of antidiuretic hormone (ADH) are elevated in patients with stroke correlating with disease severity and stress level; however, its measurement is cumbersome. ADH is derived from a larger precursor peptide along with Copeptin, which is a more stable peptide directly mirroring the production of ADH. Copeptin can be assayed readily in plasma. Early prognostic factors to predict in-hospital mortality and medium/long-term outcome in critically ill neurological patients, are helpful to guide and tailor early decisions on treatment, discharge from the intensive care unit and application of interventions to prevent deterioration of neurological functions.

We hypothesize that copeptin will improve the diagnostic accuracy to diagnose sodium imbalances as compared to routinely used markers Furthermore, we hypothesize that Copeptin will be a reliable prognostic tool, dependent or independent of sodium imbalance, to predict short-term (i.e. in-hospital) and medium-term (i.e. 3 months) clinical outcome in stroke patients.

DETAILED DESCRIPTION:
Background:

Sodium imbalance is common and an adverse prognostic factor in hospitalized patients. However, identifying the causes of sodium imbalance is challenging in clinical practice. Levels of antidiuretic hormone (ADH) are elevated in patients with stroke correlating with disease severity and stress level; however, its measurement is cumbersome. ADH is derived from a larger precursor peptide along with Copeptin, which is a more stable peptide directly mirroring the production of ADH. Copeptin can be assayed readily in plasma. Early prognostic factors to predict in-hospital mortality and medium/long-term outcome in critically ill neurological patients, are helpful to guide and tailor early decisions on treatment, discharge from the intensive care unit and application of interventions to prevent deterioration of neurological functions.

Aim: To evaluate Copeptin as a diagnostic tool in disturbances of water homeostasis and prognostic tool to predict outcome in a well-defined cohort of stroke patients and patients undergoing intracranial surgery.

Design: Prospective, observational study. Location Setting: Emergency and neurological and neurosurgical clinic of the University Hospital of Basel.

Patients: Neurological patients with ischemic and hemorrhagic stroke and patients undergoing intracranial surgery.

Intervention: After informed consent, all routinely determined baseline data will be assessed including medical history, clinical items (i.e. neurological status, volume status, pulse rate, blood pressure, weight) and laboratory items (i.e. urine / serum osmolality, electrolytes, among others). All patients will have a follow-up with clinical and laboratory assessment until the day of discharge. After 3 months, they will be followed-up by a structured telephone interview to assess outcome (mortality, morbidity, as assessed by the ranking scale and Barthel index). Copeptin will be assessed in a batch analysis upon completion of the plasma asseveration.

Variables and measurements: Baseline data on medical history and clinical items, co-morbidities and treatment procedures will be collected. This exploratory study will be conducted over a 12 month period from November 2006 to November 2007.

Study hypothesis: 1. Copeptin will improve the diagnostic accuracy to diagnose sodium imbalances as compared to routinely used markers 2. Copeptin will be a reliable prognostic tool, dependent or independent of sodium imbalance, to predict short-term (i.e. in-hospital) and medium-term (i.e. 3 months) clinical outcome in stroke patients.

Analysis: Our sample size consideration is based on the second prognostic question to predict the outcome of neurological and neurosurgical patients. To determine an optimal clinical model we will undertake a multivariable regression analysis to assess which variables are independently associated with outcome. Multiple regression models with a minimum of 10 to 15 observations per predictor variable reveal good estimates. We will evaluate 18 predictors in our multivariate analysis. Therefore, we aim to include a minimum sample size of 180 patients (for 10 observations per predictor) to 270 (for 15 observations per predictor) and a maximum sample size of 360 patients (for 20 observations per predictor).

Significance: Despite the frequent occurrence and the poor outcomes of serious disorders of sodium balance, few controlled data are available to guide the clinician. A better diagnostic approach to determine the etiology of hyponatremia should improve patient management. Copeptin as a prognostic marker in neurological and neurosurgical patients could become an innovative tool to guide early treatment decisions, discharge from the stroke unit and application of interventions.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive patients who are admitted to the emergency department with an ischemic or hemorrhagic stroke or transient ischemic attach (TIA) according to the World Health organization criteria [37] with symptom onset within the last 3 days.
2. All consecutive patients who undergo intracranial surgery due to

   * pituitary tumors
   * intracerebral hemorrhage (ICH)
   * subarachnoidal hemorrhage (SAH)
   * chronic subdural hematoma
   * head trauma with contusion cerebri
   * intracranial abcesses

Exclusion Criteria:

* Patients without informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who are admitted to the emergency department with an ischemic or hemorrhagic stroke or transient ischemic attach (TIA) according to the World Health organization criteria [37] with symptom onset within the last 3 days.
Sampling Method: Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beat Mueller, Prof, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Schweizer J, Bustamante A, Lapierre-Fetaud V, Faura J, Scherrer N, Azurmendi Gil L, Fluri F, Schutz V, Luft A, Boned S, Sanchez JC, Montaner J, Katan M. SAA (Serum Amyloid A): A Novel Predictor of Stroke-Associated Infections. Stroke. 2020 Dec;51(12):3523-3530. doi: 10.1161/STROKEAHA.120.030064. Epub 2020 Nov 9. PMID 33161846
- [Derived] De Marchis GM, Dankowski T, Konig IR, Fladt J, Fluri F, Gensicke H, Foerch C, Findling O, Kurmann R, Fischer U, Luft A, Buhl D, Engelter ST, Lyrer PA, Christ-Crain M, Arnold M, Katan M. A novel biomarker-based prognostic score in acute ischemic stroke: The CoRisk score. Neurology. 2019 Mar 26;92(13):e1517-e1525. doi: 10.1212/WNL.0000000000007177. Epub 2019 Mar 1. PMID 30824558
- [Derived] Nigro N, Wildi K, Mueller C, Schuetz P, Mueller B, Fluri F, Christ-Crain M, Katan M. BNP but Not s-cTnln is associated with cardioembolic aetiology and predicts short and long term prognosis after cerebrovascular events. PLoS One. 2014 Jul 29;9(7):e102704. doi: 10.1371/journal.pone.0102704. eCollection 2014. PMID 25072816
- [Derived] Frontzek K, Fluri F, Siemerkus J, Muller B, Gass A, Christ-Crain M, Katan M. Isolated insular strokes and plasma MR-proANP levels are associated with newly diagnosed atrial fibrillation: a pilot study. PLoS One. 2014 Mar 19;9(3):e92421. doi: 10.1371/journal.pone.0092421. eCollection 2014. PMID 24647802
- [Derived] Blum CA, Mueller C, Schuetz P, Fluri F, Trummler M, Mueller B, Katan M, Christ-Crain M. Prognostic value of dehydroepiandrosterone-sulfate and other parameters of adrenal function in acute ischemic stroke. PLoS One. 2013 May 1;8(5):e63224. doi: 10.1371/journal.pone.0063224. Print 2013. PMID 23650556
- [Derived] Zweifel C, Katan M, Schuetz P, Ernst A, Mariani L, Muller B, Christ-Crain M. Growth hormone and outcome in patients with intracerebral hemorrhage: a pilot study. Biomarkers. 2011 Sep;16(6):511-6. doi: 10.3109/1354750X.2011.599074. Epub 2011 Aug 3. PMID 21812576
- [Derived] Katan M, Fluri F, Schuetz P, Morgenthaler NG, Zweifel C, Bingisser R, Kappos L, Steck A, Engelter ST, Muller B, Christ-Crain M. Midregional pro-atrial natriuretic peptide and outcome in patients with acute ischemic stroke. J Am Coll Cardiol. 2010 Sep 21;56(13):1045-53. doi: 10.1016/j.jacc.2010.02.071. PMID 20846604
- [Derived] Urwyler SA, Schuetz P, Fluri F, Morgenthaler NG, Zweifel C, Bergmann A, Bingisser R, Kappos L, Steck A, Engelter S, Muller B, Christ-Crain M, Katan M. Prognostic value of copeptin: one-year outcome in patients with acute stroke. Stroke. 2010 Jul;41(7):1564-7. doi: 10.1161/STROKEAHA.110.584649. Epub 2010 May 27. PMID 20508186